CLINICAL TRIAL: NCT04078126
Title: A Randomized, Open-Label, Two Period Crossover, Chronic Dosing, 1-Week, Pilot Study to Assess the Efficacy and Safety of Budesonide and Formoterol Fumarate Inhalation Aerosol Administered With a Spacer Compared With Symbicort® Turbuhaler® in Subjects With Severe to Very Severe Chronic Obstructive Pulmonary Disease and Low Peak Inspiratory Flow
Brief Title: Study Comparing Dual Combination of Product (Budesonide and Formoterol) Given Via Two Different Inhalers. To See Which One Results in the Best Effect on Breathing.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D5980C00023; 2019-001801-26 (EudraCT Number)
Record Dates: First submitted 2019-09-02; First posted 2019-09-04 (Actual); Results first posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Budesonide and formoterol fumarate (MDI BFF) (Experimental): Subject treated with MDI BFF followed by washout period
  Interventions: Combination Product: BFF
- Symbicort Turbuhaler (Active Comparator): Subject treated with Symbicort followed by washout period
  Interventions: Combination Product: Symbicort Turbuhaler

INTERVENTIONS:
Combination Product: BFF — Treatment with budesonide and formoterol furmate MDI (metered-dose inhaler)
  Arms: Budesonide and formoterol fumarate (MDI BFF)
Combination Product: Symbicort Turbuhaler — Treatment with budesonide and formoterol furmate DPI (dry-powder inhaler)
  Arms: Symbicort Turbuhaler

SUMMARY:
Study comparing the same drugs as a dual combination product (budesonide and formoterol) given via two different inhalers. To see which one results in the best effect on breathing.

DETAILED DESCRIPTION:
This is a Randomized, Open-Label, Two Period Crossover, Chronic Dosing, 1-Week, Pilot Study to Assess the Efficacy and Safety of Budesonide and Formoterol Fumarate Inhalation Aerosol Administered with a Spacer Compared with Symbicort® Turbuhaler® in Subjects with Severe to Very Severe Chronic Obstructive Pulmonary Disease and Low Peak Inspiratory Flow to assess lung function

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject must be 40 to 80 years of age inclusive, at the time of signing the ICF.
2. Individuals who have a physician diagnosis of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS)
3. Require COPD maintenance therapy: all subjects must be receiving 2 or more inhaled maintenance therapies, including at least 1 long-acting bronchodilator, for the management of their COPD for at least 4 weeks prior to Visit 1.
4. A post-bronchodilator FEV1/FVC of <0.70 and post-bronchodilator FEV1 of <50% predicted normal value at Visit 2.
5. A pre-bronchodilator PIF of <50 L/min using the InCheck Inspiratory Flow Measurement Device set to Turbuhaler S resistance at Visit 2.
6. Current or former smokers with history of at least 10 pack-years of cigarette smoking.

Key Exclusion Criteria:

1. Current diagnosis of asthma, in the opinion of the Investigator.
2. Other respiratory disorders including known active tuberculosis, lung cancer, cystic fibrosis, significant bronchiectasis (high resolution CT evidence of bronchiectasis that causes repeated acute exacerbations), immune deficiency disorders, severe neurological disorders affecting control of the upper airway, sarcoidosis, idiopathic interstitial pulmonary fibrosis, primary pulmonary hypertension, or pulmonary thromboembolic disease.
3. A moderate or severe exacerbation of COPD ending within 6 weeks prior to randomization (Visit 3).
4. Need for mechanical ventilation within 3 months prior to Visit 1.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bärbel Huber, Dr., Principal Investigator — 2601; Heiner Steffen, Dr., Principal Investigator — 2602; Claus Keller, Dr., Principal Investigator — 2603; Martin Hoffmann, Dr., Principal Investigator — 2604
Locations (4):
- Germany (4):
  - Research Site, Frankfurt am Main
  - Research Site, Gauting
  - Research Site, Hanover
  - Research Site, Landsberg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Huber B, Keller C, Jenkins M, Raza A, Aurivillius M. Effect of inhaled budesonide/formoterol fumarate dihydrate delivered via two different devices on lung function in patients with COPD and low peak inspiratory flow. Ther Adv Respir Dis. 2022 Jan-Dec;16:17534666221107312. doi: 10.1177/17534666221107312. PMID 35815354
- See also: The CSP redacted. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5980C00023&attachmentIdentifier=f9e68af7-6312-4372-b1bf-35effeef648e&fileName=d5980c00023-csp-v4_Redacted_(23-Nov-2021).pdf&versionIdentifier=
- See also: the SAP redacted. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5980C00023&attachmentIdentifier=9badafff-7cec-4872-a850-18a47ba8b760&fileName=d5980C00023-sap-ed-2.1_Redacted_(23-Nov-2021).pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started recruitment in September 2019 with first subject randomized in January 2020. A total of 35 subjects were randomized at 4 study centers. The study completed in Dec 2020.
Pre-assignment Details: Subjects were randomized to an open-label, 2 period crossover study comparing Budesonide Formoterol Fumarate (BFF) Metered Dose Inhalation (MDI) administered with a spacer twice daily (BID) with Symbicort Turbuhaler BID. The subjects underwent an intervening two-week washout period where they used Berodual and Budesonide MDI BID.
Groups:
- BFF MDI/Symbicort Turbuhaler: Subject treated with Budesonide Formoterol Fumarate Metered Dose Inhalation followed by washout period and then Symbicort Turbuhaler
- Symbicort Turbuhaler/BFF MDI: Subject treated with Symbicort Turbuhaler followed by washout period and then Budesonide Formoterol Fumarate Metered Dose Inhalation
Period: Period 1
Arm/Group | BFF MDI/Symbicort Turbuhaler | Symbicort Turbuhaler/BFF MDI
Started | 18 | 17
Completed | 18 | 17
Not Completed | 0 | 0
Period: Washout
Arm/Group | BFF MDI/Symbicort Turbuhaler | Symbicort Turbuhaler/BFF MDI
Started | 18 | 17
Completed | 18 | 15
Not Completed | 0 | 2
Not completed — Study put on hold due to COVID-19 | 0 | 2
Period: Period 2
Arm/Group | BFF MDI/Symbicort Turbuhaler | Symbicort Turbuhaler/BFF MDI
Started | 18 | 15
Completed | 17 | 14
Not Completed | 1 | 1
Not completed — Study put on hold due to COVID-19 | 1 | 1

BASELINE CHARACTERISTICS:
Population: ITT Population - all subjects who were randomized to treatment
Groups:
- Overall Study: Intent-to-Treat (ITT) Population
Arm/Group | Overall Study
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] — ITT Population; mean age in years
  Years
    Mean age (SD), years | 65.8 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants] — ITT Population; Gender distribution
  Participants
    Distribution of Male/Female Participants: Female | 19
    Distribution of Male/Female Participants: Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants] — ITT Population; Race distribution
  Participants
    Race for all subjects: American Indian or Alaska Native | 0
    Race for all subjects: Asian | 0
    Race for all subjects: Native Hawaiian or Other Pacific Islander | 0
    Race for all subjects: Black or African American | 0
    Race for all subjects: White | 35
    Race for all subjects: More than one race | 0
    Race for all subjects: Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Peak Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) Within 4 Hours Post-dose Following 1 Week of Treatment
Description: Peak change from baseline in FEV1 within 4 hours post-dose was defined as the maximum of the FEV1 assessments within 4 hours post-dosing at each visit minus baseline, provided that there were at least 2 non-missing values during the first 4 hours post dose.
Time Frame: baseline and 4 hours post dose after 1 week of treatment
Population: Modified Intent-to-treat (mITT) Population included all patients who were randomized to treatment and received at least one dose of study treatment with post-baseline spirometry data from both treatment periods at Visits 4 and 6. Patients with data judged to be impacted by important protocol deviations were excluded. Patients discontinued and restarted due to the study having been put on hold for the COVID-19 pandemic used the instance of enrollment after they restarted.
Measure: Least Squares Mean (95% Confidence Interval); unit: L
Groups:
- BFF MDI: Subject treated with Budesonide Formoterol Fumarate Metered Dose Inhalation
- Symbicort Turbuhaler: Subject treated with Symbicort Turbuhaler
Arm/Group | BFF MDI | Symbicort Turbuhaler
Number analyzed (Participants) | 30 | 30
L | 0.256 [0.190 to 0.322] | 0.274 [0.208 to 0.340]
Statistical Analysis 1: Comparison: BFF MDI vs Symbicort Turbuhaler; Test type: Other; p = 0.3450, ANCOVA; Mean Difference (Final Values) = -0.017, 95% CI 2-sided [-0.054 to 0.020], Standard Error of Mean 0.0179

2. Secondary Outcome: Area Under the Curve for Change From Baseline in FEV1 From Area Under the Curve 0 to 4 Hours (AUC0-4 h) Following 1 Week of Treatment
Description: FEV1 AUC0-4 was calculated using the trapezoidal rule and was normalized by dividing by the time in hours from dosing to the last measurement included (typically 4 hours).
Time Frame: baseline and 4 hours post dose after 1 week of treatment
Population: mITT Population included all patients who were randomized to treatment and received at least one dose of study treatment with post-baseline spirometry data from both treatment periods at Visits 4 and 6. Patients with data judged to be impacted by important protocol deviations were excluded. Patients discontinued and restarted due to the study having been put on hold for the COVID-19 pandemic used the instance of enrollment after they restarted.
Measure: Least Squares Mean (95% Confidence Interval); unit: L
Arm/Group | BFF MDI | Symbicort Turbuhaler
Number analyzed (Participants) | 30 | 30
L | 0.194 [0.133 to 0.254] | 0.210 [0.149 to 0.271]
Statistical Analysis 1: Comparison: BFF MDI vs Symbicort Turbuhaler; Test type: Other; p = 0.3675, ANCOVA; Mean Difference (Final Values) = -0.017, 95% CI 2-sided [-0.054 to 0.021], Standard Error of Mean 0.0183

3. Secondary Outcome: Change From Baseline in Pre-dose FEV1 Following 1 Week of Treatment
Description: Change from baseline in pre-dose FEV1 following 1 week of treatment was defined as the 45-minute pre-dose value following 1 week of treatment minus baseline.
Time Frame: baseline and after 1 week of treatment
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: L
Arm/Group | BFF MDI | Symbicort Turbuhaler
Number analyzed (Participants) | 30 | 30
L | 0.081 [0.030 to 0.131] | 0.087 [0.037 to 0.137]
Statistical Analysis 1: Comparison: BFF MDI vs Symbicort Turbuhaler; Test type: Other; p = 0.7563, ANCOVA; Mean Difference (Final Values) = -0.006, 95% CI 2-sided [-0.047 to 0.034], Standard Error of Mean 0.0199

4. Secondary Outcome: Change From Baseline in 2-hour Post-dose Inspiratory Capacity (IC) Following 1 Week of Treatment
Description: Change from baseline in 2-hour post-dose IC following 1 week of treatment was defined as the 2-hour post-dose assessment of IC following 1 week of treatment minus baseline IC.
Time Frame: baseline and 2 hours post dose after 1 week of treatment
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: L
Arm/Group | BFF MDI | Symbicort Turbuhaler
Number analyzed (Participants) | 30 | 30
L | 0.379 [0.242 to 0.517] | 0.411 [0.275 to 0.548]
Statistical Analysis 1: Comparison: BFF MDI vs Symbicort Turbuhaler; Test type: Other; p = 0.5419, ANCOVA; Mean Difference (Final Values) = -0.032, 95% CI 2-sided [-0.139 to 0.075], Standard Error of Mean 0.0521

5. Secondary Outcome: Change From Baseline in Pre-dose Peak Inspiratory Flow (PIF; InCheck Device Set to no Resistance) Following 1 Week of Treatment
Description: Change from baseline in pre-dose PIF (InCheck device set to no resistance) following 1 week of treatment was defined as the pre-dose PIF (InCheck device set to no resistance) following 1 week of treatment minus baseline PIF. (The InCheck Inspiratory Flow Measurement Device is an inhalation airflow meter that may be set to various resistances similar to marketed inhaler products. For this measurement, the device was set to no resistance.)
Time Frame: baseline and after 1 week of treatment
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | BFF MDI | Symbicort Turbuhaler
Number analyzed (Participants) | 30 | 30
L/min | 1.50 [-2.26 to 5.27] | 5.11 [1.34 to 8.88]
Statistical Analysis 1: Comparison: BFF MDI vs Symbicort Turbuhaler; Test type: Other; p = 0.1337, ANCOVA; Mean Difference (Final Values) = -3.60, 95% CI 2-sided [-8.39 to 1.18], Standard Error of Mean 2.334

6. Secondary Outcome: Change From Baseline in Pre-dose PIF (Resistance Set Equal to Turbuhaler S) Following 1 Week of Treatment
Description: Change from baseline in pre-dose PIF (resistance set equal to Turbuhaler S) following 1 week of treatment was defined as the pre-dose PIF (resistance set equal to Turbuhaler S) following 1 week of treatment minus baseline PIF. (The InCheck Inspiratory Flow Measurement Device is an inhalation airflow meter that may be set to various resistances similar to marketed inhaler products. For this measurement, the device was set to resistance equal to the product Turbuhaler S.)
Time Frame: baseline and after 1 week of treatment
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | BFF MDI | Symbicort Turbuhaler
Number analyzed (Participants) | 30 | 30
L/min | 1.13 [-0.78 to 3.03] | 3.82 [1.91 to 5.72]
Statistical Analysis 1: Comparison: BFF MDI vs Symbicort Turbuhaler; Test type: Other; p = 0.0431, ANCOVA; Mean Difference (Final Values) = -2.69, 95% CI 2-sided [-5.29 to -0.09], Standard Error of Mean 1.269

7. Secondary Outcome: Change From Baseline in Pre-dose PIF (Resistance Set Equal to ELLIPTA) Following 1 Week of Treatment
Description: Change from baseline in pre-dose PIF (resistance set equal to ELLIPTA) following 1 week of treatment was defined as the pre-dose PIF (resistance set equal to ELLIPTA) following 1 week of treatment minus baseline PIF. (The InCheck Inspiratory Flow Measurement Device is an inhalation airflow meter that may be set to various resistances similar to marketed inhaler products. For this measurement, the device was set to resistance equal to the product ELLIPTA.)
Time Frame: baseline and after 1 week of treatment
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | BFF MDI | Symbicort Turbuhaler
Number analyzed (Participants) | 30 | 30
L/min | 1.21 [-1.15 to 3.56] | 2.74 [0.39 to 5.09]
Statistical Analysis 1: Comparison: BFF MDI vs Symbicort Turbuhaler; Test type: Other; p = 0.3625, ANCOVA; Mean Difference (Final Values) = -1.53, 95% CI 2-sided [-4.87 to 1.81], Standard Error of Mean 1.667

8. Secondary Outcome: Change From Baseline in 2-hour Post-dose FEV1 Following the First Dose
Description: Change from baseline in 2-hour post-dose FEV1 following the 1st dose of treatment was defined as the 2-hour post-dose assessment of FEV1 following the 1st dose of treatment (Visit 3 or 5) minus baseline FEV1.
Time Frame: baseline and 2 hours post dose after the first dose of treatment
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: L
Arm/Group | BFF MDI | Symbicort Turbuhaler
Number analyzed (Participants) | 30 | 30
L | 0.136 [0.100 to 0.173] | 0.093 [0.057 to 0.130]
Statistical Analysis 1: Comparison: BFF MDI vs Symbicort Turbuhaler; Test type: Other; p = 0.0375, ANCOVA; Mean Difference (Final Values) = 0.043, 95% CI 2-sided [0.003 to 0.084], Standard Error of Mean 0.0198

9. Secondary Outcome: Change From Baseline in 2-hour Post-dose IC Following the First Dose
Description: Change from baseline in 2-hour post-dose IC following the 1st dose of treatment was defined as the 2-hour post-dose assessment of IC following the 1st dose of treatment (Visit 3 or 5) minus baseline IC.
Time Frame: baseline and 2 hours post dose after the first dose of treatment
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: L
Arm/Group | BFF MDI | Symbicort Turbuhaler
Number analyzed (Participants) | 28 | 30
L | 0.264 [0.164 to 0.363] | 0.258 [0.161 to 0.356]
Statistical Analysis 1: Comparison: BFF MDI vs Symbicort Turbuhaler; Test type: Other; p = 0.9089, ANCOVA; Mean Difference (Final Values) = 0.005, 95% CI 2-sided [-0.086 to 0.096], Standard Error of Mean 0.0443

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were monitored/assessed from Randomization throughout the Treatment Period and including the washout and follow-up periods, a maximum of 6 weeks. Serious adverse events were recorded from the time of signing of the informed consent, through Run-in, Treatment Period, including washout, and follow-up period, a maximum of 9 weeks.
Description: The Safety Population was defined as all subjects who were randomized to treatment and received at least one dose of study treatment. Subjects were analyzed according to the treatment actually received.
Arm/Group | BFF MDI | Symbicort Turbuhaler
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/35
Other Adverse Events (participants affected / at risk) | 1/33 | 1/35
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BFF MDI (N=33) | Symbicort Turbuhaler (N=35)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT04078126/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT04078126/SAP_001.pdf